CLINICAL TRIAL: NCT05739331
Title: Automatic Segmentation of Mediastinal Lymph Nodes and Blood Vessels in Endobronchial Ultrasound (EBUS) Images Using a Deep Neural Network
Brief Title: Augmented Endobronchial Ultrasound (EBUS-TBNA) With Artificial Intelligence
Status: Recruiting | Type: Observational
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: Helse Nord-Trøndelag HF (Other); SINTEF Health Research (Other)
Responsible Party: Sponsor
Other Study IDs: 240245
Record Dates: First submitted 2023-02-13; First posted 2023-02-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-06

CONDITIONS: Artificial Intelligence; Endobronchial Ultrasound; Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: machine learning algorithm — Machine learning algorithm run on EBUS images for real-time labelling of mediastinal lymph nodes and lymph node level

SUMMARY:
To evaluate the usefulness of Deep neural network (DNN) in the evaluation of mediastinal and hilar lymph nodes with Endobronchial ultrasound (EBUS). The study will explore the feasibility of DNN to identify lymph nodes and blood vessel examined with EBUS.

DETAILED DESCRIPTION:
Multi-center prospective feasibility study. The DNN model will be trained on ultrasound images with annotation to identifies lymph nodes and blood vessels examined with EBUS. The ability of the DNN to segment lymph nodes and vessels based on postoperative processing and static EBUS images will be evaluated in the first part of the study. In the second part of the study Real-time use of DNN in EBUS procedure will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Subjects referred to thoracic department in any of the participating hospitals with undiagnosed enlarged mediastinal and hilar lymph nodes.
* Subjects have to be ≥ 18 years of age

Exclusion Criteria:

* Pregnancy
* Any patient that the Investigator feels is not appropriate for this study for any reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patents with undiagnosed enlarged mediastinal and hilar lymph nodes who have been recommended for Endobronchial ultrasound transbronchial needle aspiration (EBUS-TBNA).
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Capability | 8 months
  To explore if Deep neural network (DNN) has capability to segment lymph nodes and blood vessels from EBUS images

SECONDARY OUTCOMES:
Precision | 2 months
  The precision the DNN has for detecting lymph nodes and blood vessels. Measured both per voxel in the EBUS images and per annotated structure (a structure is counted as detected if at least 50% of its annotated pixels are identified by the DNN).
Sensitivity | 2 months
  True positive rate. Correctly detected lymph nodes/blood vessel over total lymph nodes/blood vessel. Measured per pixel in the EBUS images
Specificity | 2 months
  Specificity = (True Negative)/(True Negative + False Positive). Measured per pixel in the EBUS images.
Dice similarity coefficient | 2 months
  Measures the similarity between two sets of data: Annotated by pulmonologist vs DNN.
Run-time | 2 months
  Is the run-time sufficiently low for real-time analysis during EBUS?
Adverse events | 48 hours
  Procedure related adverse events or unexpected incidents registered

CONTACTS AND LOCATIONS:
Overall Officials: Øivind Rognmo, Dr.philos, Study Director — Norwegian University of Science and Technology
Locations (2):
- Norway (2):
  - Department of Pulmonology, Levanger Hospital, North Trøndelag Hospital Trust, Levanger
  - Department of Thoracic Medicine, St Olavs Hospital, Trondheim